CLINICAL TRIAL: NCT03816592
Title: Opioid Free Anaesthesia in Cardiac Surgery With Cardiopulmonary Bypas
Brief Title: Opioid Free Anaesthesia in Cardiac Surgery With Cardiopulmonary Bypass
Acronym: OFACAR 1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GUINOT 2019
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Opioid Free Anaesthesia; Opioid Anaesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Opioid free anaesthesia: patient anesthtesized with lidocaine, ketamine and dexamethasone
  Interventions: Procedure: Opioid free anaesthesia
- Opioid anaesthesia: patients anesthetized with sufentanil ketamine and dexamethasone
  Interventions: Procedure: Opioid anaesthesia

INTERVENTIONS:
Procedure: Opioid free anaesthesia — patient anesthtesized with lidocaine, ketamine and dexamethasone
  Groups: Opioid free anaesthesia
Procedure: Opioid anaesthesia — patients anesthetized with sufentanil ketamine and dexamethasone
  Groups: Opioid anaesthesia

SUMMARY:
Since the 1990s, the concept of anesthesia without morphine (OFA) has been developed. The principle is based on the fact that in a sleeping patient a sympathetic reaction marked by hemodynamic changes does not reflect a painful phenomenon, that a painful phenomenon in a sleeping patient is not memorized, that hormonal stress, sympathetic reaction and inflammatory reaction can be controlled by therapeutic classes other than a morphine agent. This therapeutic management would avoid the side effects associated with the use of morphine. In cardiac surgery, no studies have evaluated the effect of an OFA on morphine consumption and on a post-operative composite endpoint. Lidocaine was only studied in the context of cardioprotection and neuroprotection. Studies found a cardioprotective effect with a decrease in episodes of rhythmic disorders, and neuroprotective with a non-constant improvement in postoperative cognitive functions, but all these studies were performed during opioid anaesthesia (opioid agent use)/ The purpose of our study is to demonstrate that general anesthesia without opioid (OFA) is associated with a decrease in post-operative morphine consumption and an improvement in the patient's post-operative well-being (complications, confusion, vigilance, length of stay).

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* patient with chronic analgesia treatment
* patient on antidepressive therapy
* gabapentin use
* preoperative cognitive dysfunction
* patient treated with zyvoxid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgical
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Day 2
  Total morphine consumption over the first 48 post operative hours in milligrammes
Complications | Day 7
  composite end point of post operative complications (cardiac, neurological, renal, respiratory)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Guinot PG, Spitz A, Berthoud V, Ellouze O, Missaoui A, Constandache T, Grosjean S, Radhouani M, Anciaux JB, Parthiot JP, Merle JP, Nowobilski N, Nguyen M, Bouhemad B. Effect of opioid-free anaesthesia on post-operative period in cardiac surgery: a retrospective matched case-control study. BMC Anesthesiol. 2019 Jul 31;19(1):136. doi: 10.1186/s12871-019-0802-y. PMID 31366330